CLINICAL TRIAL: NCT06682000
Title: A Multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of DWC202404 and DWC202314 Combination Therapy in Patients With Essential Hypertension Inadequately Controlled on DWC202404 Monotherapy
Brief Title: Efficacy and Safety of DWC202404 and DWC202314 in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1621301
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Essential Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWC202404 + DWC202314 (Experimental)
  Interventions: Drug: DWC202404, DWC202314
- DWC202404 + DWC202314P (Placebo Comparator)
  Interventions: Drug: DWC202404, DWC202314P

INTERVENTIONS:
Drug: DWC202404, DWC202314 — - 2 tablet, Oral, Once a day
  Arms: DWC202404 + DWC202314
Drug: DWC202404, DWC202314P — - 2 tablet, Oral, Once a day
  Arms: DWC202404 + DWC202314P

SUMMARY:
A Multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of DWC202404 and DWC202314 Combination Therapy in Patients with Essential Hypertension Inadequately Controlled on DWC202404 Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Average systolic blood pressure (MSSBP) measured at the time of screening meet the following criteria (a) If anti-hypertensive drugs are not being administered: 140 mmHg ≤ MSSBP < 180 mmHg (b) If anti-hypertensive drugs are being administered: 130 mmHg ≤ MSSBP < 180 mmHg

Exclusion Criteria:

* If the blood pressure measured at the time of screening and randomization is MSDBP ≥ 110 mmHg
* Those whose blood pressure differences measured on both arms at the time of screening are MSSBP ≥ 20 mmHg and MSDBP ≥ 10 mmHg

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change of MSSBP (Mean Sitting Systolic Blood Pressure) based on baseline | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea